CLINICAL TRIAL: NCT05820737
Title: A Randomized, Double Blind, Placebo Controlled, Parallel Group Study to Assess the Gut Health Effects of Heat-killed Post-biotics EF2001 & beLP1 in Overweight and Obese Adults
Brief Title: A Study to Assess the Gut Health Effects of Heat-killed Post-biotics in Overweight and Obese Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vedic Lifesciences Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: BR/221101/EFLP/GH
Record Dates: First submitted 2023-04-06; First posted 2023-04-20 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2024-01

CONDITIONS: Gastrointestinal Dysfunction

STUDY DESIGN:
Intervention Model Description: Randomized, parallel group, placebo controlled trial
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): 1 capsule to be consumed once a day
  Interventions: Dietary Supplement: Placebo
- EF2001 (Active Comparator): 1 capsule to be consumed once a day
  Interventions: Dietary Supplement: EF2001
- beLP1 (Active Comparator): 1 capsule to be consumed once a day
  Interventions: Dietary Supplement: beLP1

INTERVENTIONS:
Dietary Supplement: EF2001 — One capsule to be consumed once a day
  Arms: EF2001
Dietary Supplement: beLP1 — One capsule to be consumed once a day
  Arms: beLP1
Dietary Supplement: Placebo — One capsule to be consumed once a day
  Arms: Placebo

SUMMARY:
The present study is a randomized, double-blind (Double dummy), placebo-controlled, parallel-group study to assess the gut health effects of heat-killed post biotics in overweight and obese individuals

ELIGIBILITY:
Inclusion Criteria:

* Male and female individuals with the age ≥18 and ≤45 years with active lifestyle, moderate physical activity level as per International Physical Activity Questionnaire - Short Form (IPAQ-SF - SF)
* BMI of ≥ 25 - ≤ 35 kg/m2
* Individuals with liver & renal function test values as defined below:

  1. Individuals with ALT, AST values ≤ 2 times of the upper limit of normal (ULN).
  2. Individuals with creatinine values ≤ 1.5 times of the upper limit of normal (ULN).
  3. Individuals with ALP values ≥ 38 and ≤ 126 U/L
* Having at least two of the following five metabolic risk factors:

  1. Waist circumference > 102 cm (40 inches) for men and > 88 cm (35 inches) for women
  2. Fasting triglycerides >150 mg/dL and < 300 mg/dl
  3. Blood pressure ≥130 mm Hg (Systolic Blood Pressure) and/or ≥85 mm Hg (Diastolic Blood Pressure)
  4. Fasting blood glucose ≥ 100 mg/ dl
  5. Fasting HDL cholesterol level less than 40 mg/dl (men) or 50 mg/dl (women)
* History of mild to moderate gastrointestinal discomfort for at least last three months
* Individuals experiencing moderate-intensity gastrointestinal symptoms, evaluated based on the combined scores of two GSRS domains (dyspeptic syndrome and bowel dysfunction), falling within the range of ≥ 15 and ≤ 29 over the past two weeks. (The highest score out of two weeks' GSRS scores will be taken into consideration for the study)
* Willing to complete all study procedures including study-related questionnaires and comply with study requirements.
* Willing to abstain from other supplements or medication.
* Ready to give voluntary, written, informed consent to participate in the study
* No prohibited antibiotic usage within the last 30 days.
* History of stable weight over the last 6 months (<10% change)
* Willing to maintain current dietary and exercise habits, aside from any changes to be made per the study exercise protocol

Randomization Criteria:

* Two weeks of run - in period for weight stability (Weight instability defined as > 2 kg of weight gain or loss over 2 weeks of run-in period)
* GSRS scores not less than that reported at screening. (The highest score out of two weeks' GSRS scores will be taken into consideration for the study)
* Both the weekly at-home diaries for GSRS should be available
* 80% compliance to the run-in medication

Exclusion Criteria:

* Individual who smokes and consumes tobacco regularly.
* Presence of unstable, acutely symptomatic, or life-limiting illness.

  * Individuals diagnosed with diabetes and are on active medication
  * FBG > 125 mg/dl
  * Individuals diagnosed with hypertension and are on active medication.
  * Individuals with uncontrolled hypertension with systolic blood pressure ≥150 and/or diastolic blood pressure ≥100 mm Hg.
* Individuals with neurological conditions causing functional or cognitive impairments.

  * Individuals with a history or presence of clinically significant renal, hepatic, endocrine, biliary, gastrointestinal, pancreatic or neurologic disorders that, in the judgment of the Investigator, would interfere with the subject's ability to provide informed consent, comply with the study protocol (which might confound the interpretation of the study results), or put the subject at undue risk.
  * Individuals under use of any psychotropic medication within four weeks of screening and throughout the study
* Individual under use of antibiotics or signs of active systemic infection at the time of screening. Treatment visits will be rescheduled to allow the subject to wash off the antibiotic for at least five days prior to any test visit
* Individual states they regularly consume supplemental enzymes and are unwilling to stop at least one week prior to screening and throughout the study. Supplemental enzymes may include standalone enzyme supplements, probiotic supplements with enzymes, and any medications containing enzymes.

  * Individuals states they regularly consume probiotic supplements and are unwilling to stop at least one week prior to screening and throughout the study. Supplemental probiotics may include standalone probiotic supplements, vitamins with probiotics, and any foods supplemented with probiotics
  * Exposure to any non-registered drug product within 3 months prior to the screening visit.
  * Unable/unwillingness to complete study specific diaries (digital/paper-based).
  * Current use of the following medications: monoamine oxidase inhibitors, prescription or herbal weight loss medications/ dietary supplement.
  * Females who are pregnant/planning to be pregnant/lactating or taking any oral contraceptives.
  * Individual who reports alcohol intake as average of 3 or more servings per day 18. Individuals with thyroid dysfunction as assessed by TSH ≤ 0.4 or ≥ 4.3 mIU/L.
* Individuals state they have an allergy or intolerance to any ingredient in the study product or test meal.

  * Individual is deemed unsuitable for study based upon study physician assessment.
  * Individual is taking part in another clinical trial

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 155 (Actual)
Dates: Start 2024-04-14 (Actual); Primary Completion 2025-03-24 (Actual); Study Completion 2025-03-24 (Actual)

PRIMARY OUTCOMES:
To assess efficacy of the Post-biotics on Gastrointestinal Symptom Rating Scale (GSRS) from baseline. | Day 42 and Day 84
  Questions are to be rated on a Likert scale ranging from no discomfort at all (0) to very severe discomfort (3). A total score is calculated by summing the ratings provided on all questions. The questionnaire has 18 items - epigastric pain, colicky pain, dull pain, undefined pain, heartburn, acid regurgitation, sucking sensation, nausea and vomiting, borborygmus, abdominal distension, eructation, increased flatus, decreased passage of stools, increased passage of stools, loose stools, hard stools, urgent need for defecation and feeling of incomplete evacuation

SECONDARY OUTCOMES:
To assess the impact of the IP from baseline as compared to placebo on Body Composition using Dual Energy X-ray Absorptiometry scan (DEXA).. | Day 42 and Day 84
  The overall body composition (Lean Body Mass, Body Fat percent, Fat Free Mass, android and gynoid fat) will be evaluated using Dual Energy X-ray Absorptiometry scan (DEXA).
To assess the impact of the IP from baseline as compared to Gut permeability by assessing the levels of Lipopolysaccharide Binding Protein (LBP). | Day 42 and Day 84
  The amount of the LBP will be calculated based on the standard curve. A study demonstrated an average of 7.8 μg/mL of LBP in obese individuals and 6 μg/mL in normal weight individuals.
To assess the impact of the IP from baseline as compared to placebo on Homeostasis Model Assessment-Estimated Insulin Resistance (HOMA-IR) | Day 42 and Day 84
  HOMA-IR = (Fasting glucose × Insulin levels) ÷ 40 In a clinical study, subjects without metabolic syndrome exhibited a HOMA-IR value of 2.39, whereas obese subjects showed a higher HOMA-IR of 4.04.
To assess the impact of the IP from baseline as compared to placebo on Immunomodulation using INF-γ | Day 42 and Day 84
  In the current study, the impact of the heat killed postbiotics will be evaluated in enhancing the immune-modulatory characteristics in individuals under metabolic stress
To assess the impact of the IP from baseline as compared to placebo on Cytokine levels like IL-6. | Day 42 and Day 84
  IL-6 may be considered as a significant prognostic indicator of risk of any metabolic disorder.
To assess the impact of the IP from baseline as compared to placebo on Inflammation by assessing the levels of Tumor necrosis factor -alpha (TNF - α) | Day 42 and Day 84
  TNF levels were elevated in adipose tissue in obese and insulin-resistant rodents and suggested that TNF had a role in mediating insulin resistance
To assess the impact of the IP from baseline as compared to placebo on Lipid profile: Total cholesterol, Triglyceride, HDL, LDL. | Day 42 and Day 84
  The Lipid Profile will be performed on Roche cobas, Desirable cholesterol level is < 5.17 mmol/L (< 200 mg/dL). Desirable HDL level is > 1.68 mmol/L (> 65 mg/dL) in females & > 1.45 mmol/L (> 55 mg/dL) in males. Normal range of triglycerides is < 1.70 mmol/L (< 150 mg/dL)
To assess the impact of the IP from baseline on Perceived Stress Scale (PSS) | Day 42 and Day 84
  Perceived Stress Scale (PSS). Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress.
To assess the impact of the IP from baseline as compared to placebo on Quality of life using Digestive Associated Quality of Life Questionnaire. | Day 42 and Day 84
  Quality of life using Digestive Associated Quality of Life Questionnaire., The total score represents the sum of the responses to the 9 statements with possible scores ranging from 0 to 9. A higher score indicates a lower (worse) digestion-associated QOL.
To assess the impact of the IP on change in the following parameters baseline on Short Chain Fatty Acids (SCFA) | Day 84
  Short Chain Fatty Acids (SCFA)
To assess the impact of the IP on change in the following parameters from baseline on Humoral response as assessed by Th1/Th2 in plasma. | Day 84
  Th1 cells secrete the cytokine interferon-gamma and activate inflammatory pathways mainly via macrophage activation .Th2 cells secrete cytokines interleukin-4 and -5 that upregulate antibody formation via B cells, mast cells, eosinophils, and other pathways. Th1 and Th2 cells can cross-inhibit each other
To assess the impact of the IP on change in the following parameters from baseline on Gut microbiome diversity using metagenome NGS sequencing of the fecal samples. | Day 84
  Gut microbiome diversity using metagenome NGS sequencing of the fecal samples.

CONTACTS AND LOCATIONS:
Locations (9):
- India (9):
  - Dr. KotharisDigestive andLiver care, Pune, Maharashta
  - AIIMS Hospital, Dombivali, Maharashtra
  - Ramesh Dargad Clinic, Mumbai, Maharashtra
  - Sarthak Health Clinic., Nashik, Maharashtra
  - Surya Multispeciality hospita, Nashik, Maharashtra
  - Dr. Thakare superspeaciality clinic, Nashik, Maharashtra
  - Life care Hospital, Nashik, Maharashtra
  - Metabol, Ghātkopar
  - Dhanwantari Hospita, Pune

IPD SHARING:
Plan to Share IPD: Undecided